CLINICAL TRIAL: NCT02931708
Title: Diaphragmatic Functional Electrical Stimulation in Heart Failure Patients: Uncontrolled Clinical Trial
Brief Title: Diaphragmatic Functional Electrical Stimulation in Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, PhD, Federal University of Health Science of Porto Alegre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFESHF
Record Dates: First submitted 2016-09-01; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Diaphragm; Electrical Stimulation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DFES group (Experimental): Diaphragm Functional Electrical Stimulation:
  Each session will last 30 minutes. The parameters selected in the stimulator will be: 80 Hz frequency, 0.4 ms pulse, rise 1s, 1s time on, decay 2s, 1s time off, intensity as patient tolerance.
  The patient will be positioned supine, headboard 30º, knees extended. Furthermore, the electrodes used to perform the electrical stimulation will be adhesive, disposable and hypoallergenic. These will be placed at sixth, seventh and eighth intercostal spaces, axiliar medium line and paraxiphoid both chest sides.
  Interventions: Other: Diaphragm functional electrical stimulation

INTERVENTIONS:
Other: Diaphragm functional electrical stimulation — Functional electrical stimulation: 80 Hz frequency, 0.4 ms pulse, rise 1s, 1s time on, decay 2s, 1s time off, intensity as patient tolerance

SUMMARY:
Heart failure is an incapacity to provide adequate blood flow to the others organs, such as brain, liver and kidney. The patients presents weakness and fatigue of inspiratory muscles, mainly diaphragm muscle, that contributes to dyspnoea and limited physical capacity in this patients.

Some methods are being studied to decrease the diaphragm weakness. The diaphragm functional eletrical stimulation is a new technique, which has been studied to improve the respiratory muscle strength. Then, the aim of this study is to assess the effects of diaphragm functional electrical stimulation (FES) on respiratory muscle strength and muscle architecture of patients with heart failure.

For this the following assessments will be performed before and after stimulation: manovacuometry to verify the maximum inspiratory pressure and maximum expiratory pressure; and ultrasonography to assess muscle architecture.

The subjects will be selected by the decompensation in heart failure, with the adequate elegibility criteria. This study have no control group, because this technique has been little researched and could be unethical with the patient who won't receive this treatment.

The subjetcs of this research will receive the diaphragm functional electrical stimulation twice of day for consecutive five days or until the hospital discharge.

Expected results at the end of the protocol with Diaphragm Functional Electrical Stimulation are: to improve respiratory muscle strength; to correlate with diaphragm muscle arquiteture.

DETAILED DESCRIPTION:
The research will be developed in the São Francisco Hospital, of Santa Casa de Misericordia de Porto Alegre. After the selection of patients for eligibility criteria they will be evaluated, and subsequently the patients in will be trained twice of day for five days or until hospital discharge. Will be use an electric current called functional electrical stimulation through the stimulator device NEURODYN II, IBRAMED mark, Amparo, São Paulo, Brazil.

Each session will last 30 minutes. The parameters selected in the stimulator will be: 80 Hz frequency, 0.4 ms pulse, rise 1s, 1s time on, decay 2s, 1s time off, intensity as patient tolerance.

The patient will be positioned supine, headboard 30º, knees extended. Furthermore, the electrodes used to perform the electrical stimulation will be adhesive, disposable and hypoallergenic. These will be placed at sixth, seventh and eighth intercostal spaces, axiliar medium line and paraxiphoid both chest sides.

At the end of follow-up, will be compared the data of before and after interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure, being admited at the hospital for decompensation of the disease

Exclusion Criteria:

* Cognitive impairment that prevents conducting evaluations, as well as inability to understand and sign the informed consent form;
* Epidermal lesions at the site of application and/or intolerance stimulator and/or skin sensitivity change;
* Use pacemaker, cardiac resynchronization and/or implantable cardioverter defibrillator;
* Body mass index >40Kg/m²

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength assessed by manovacuometry | Five days or until hospital discharge
  Respiratory muscle strength assessed by manovacuometry

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre
Locations (1):
- Irmandade Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes